CLINICAL TRIAL: NCT03852199
Title: A Validation Study of Force Sense Measurement With a New Instrument
Brief Title: A Validation Study of Force Sense Measurement
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ceyhun Turkmen, Research Assistant, Hacettepe University
Other Study IDs: GO 18/932
Record Dates: First submitted 2019-02-19; First posted 2019-02-25 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Knee Injuries; Proprioceptive Disorders
Keywords: force sense; knee joint; proprioception; sphygmomanometer; surface EMG
MeSH Terms: conditions — Knee Injuries; Somatosensory Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Case Group: Our study was performed with 30 healthy individuals at Hacettepe University, Faculty of Physical Therapy and Rehabilitation. The FS of the knee joint was measured with a Pressure Biofeedback Device (Stabilizer ™, Chattanooga Group Inc., Chattanooga, TN), a device similar to a sphygmomanometer. To correlate the outcomes of biofeedback device, simultaneously, a surface electromyography (EMG) data of M. Quadriceps femoris muscle activation levels from the individuals were recorded.
  Interventions: Other: Test protocol for proprioceptive force sense in case group

INTERVENTIONS:
Other: Test protocol for proprioceptive force sense in case group — * The FS in the knee region was measured by the pressure, biofeedback device (Stabilizer ™, Chattanooga Group Inc., Chattanooga, TN).
  * Surface EMG device (Noraxon USA, Inc., Scottsdale, AZ) was used to measure activation levels of M. Vastus Medialis Obliquus (VMO), M. Vastus Lateralis (VL) and M. Rectus Femoris (RF) muscles. Due to the characteristics of the Bipolar Ag/AgCl surface electrodes, the distance between the electrodes was set to 1 cm and the electrode width to 2 cm. The electrode placement was determined according to the SENIAM (Surface ElectroMyoGraphy for the Non-Invasive Assessment of Muscles) criteria.

SUMMARY:
The term proprioception was first introduced by Sherrington in 1906, who described it as a type of feedback from the limbs to the central nervous system. Based on the early descriptions by Sherrington and others, the contemporary terms of joint position sense (JPS), kinaesthesia (perception of active and passive motion), and sense of tension or force sense are considered sub modalities of proprioception.

For the extremity joints, goniometers (universal, bubble, digital) can also be used to measure active JPS. Depending on the device used and the extremity joint measured, reliability and measurement error of active movement goniometry can range widely and this should be carefully considered if goniometry is used to measure active JPS of extremity joints. Kinesthesia, can be measured by calculating the passive motion detection threshold of individuals.

The force sense (FS), commonly assessed using force reproduction, has also been used as a measure of proprioception. Assessing force reproduction by limb matching involves the use of a reference force, usually determined as a percentage of a Maximal Voluntary Isometric Contraction (MVIC), and attempting to replicate that force.

Proprioception can be decreased in those who suffer from knee injury. Because patients with severe degenerative joint disease often require total knee arthroplasty to relieve pain, improve stability, and restore function. Due to problems such as oedema, immobilization and subjective pain after surgery, it is difficult to evaluate proprioception with joint repositioning method. In such cases, the assessment of FS could be of particular interest in the knee region. FS can also be measured by the accuracy of reproducing a specific target force. For example, the pressure biofeedback device (PBD) used for assessing the cranio-cervical flexion test could be considered a method of assessing force sense in the cervical spine. The ability to hold steadily or the accuracy in achieving and maintaining a desired pressure can be used. However, for the knee region, there is no method to measure the force sense via a device that can be used in clinical practice.

The aim of this study was to establish a method for measuring FS that could be applied quickly and practically in the clinic, and to correlate the outcomes with surface electromyographic (EMG) muscle activation levels from M. Quadriceps femoris to demonstrate the applicability and objectivity of this method.

ELIGIBILITY:
Inclusion Criteria:

* without chronic knee problems
* without chronic neurologic problems
* without chronic rheumatological problems
* without cognitive problems

Exclusion Criteria:

* Osteoporosis

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy individuals without chronic knee problems were included in the study.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Measurement of force sensations in mmHg with "Pressure Biofeedback Device" Measurement of Force Sense in mmHg with "Pressure Biofeedback Device" | Participants are evaluated only once in 45 minutes.
  First, the participants were positioned on the exercise bed. Then, the pressure biofeedback device was placed under the knee joint on the dominant lower extremity side and the cuff was inflated to a pressure of 20 mmHg. Before the measurement, the participants were told to press their knees to the ground and thus to bring the M.Quadriceps femoris into maximum isometric contraction. 50% and 65% of this maximum value obtained for each individual were recorded as reference values for measuring the force sense error of knee region.

CONTACTS AND LOCATIONS:
Locations (1):
- Ceyhun Türkmen, Ankara, Altindag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided